CLINICAL TRIAL: NCT02050334
Title: Protocol CC100A CC100: Safety and Tolerability of Single Doses
Brief Title: CC100: Safety and Tolerability of Single Doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chemigen, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CC100A
Record Dates: First submitted 2014-01-29; First posted 2014-01-30 (Estimated); Results first posted 2015-04-29 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: Phase 1; Healthy Volunteer; Safety; Healthy Volunteer Safety Study

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CC100 (3 single doses) (Experimental): CC100 (3 single increasing doses by mouth). Dosing will occur every 2 to 7 days for a study duration of 5 to 15 days from the 1st dose.
  Interventions: Drug: CC100
- CC100 (2 single doses) & placebo(1 dose) (Experimental): CC100 (2 single increasing doses by mouth) and placebo (1 single dose by mouth). Dosing will occur every 2 to 7 days for a study duration of 5 to 15 days from the 1st dose.
  Interventions: Drug: CC100; Drug: Placebo

INTERVENTIONS:
Drug: CC100 — CC100 reconstituted in diluent
  Other Names: synthetic caffeic acid phenethylester
Drug: Placebo — Diluent. Amount to match CC100 dose.
  Other Names: Inactive vehicle
  Arms: CC100 (2 single doses) & placebo(1 dose)

SUMMARY:
The purpose of this study is to see if CC100, given by mouth, is safe and is tolerated in increasing doses. How long the drug remains in the body will also be calculated.

DETAILED DESCRIPTION:
Approximately 18 healthy subjects will be randomized to receive by mouth either 3 single increasing doses of CC100 or 1 dose of placebo and 2 increasing doses of CC100. Dosing will occur every 2 to 7 days for a study duration of 5 to 15 days from the 1st dose. Subjects are required to stay in the Clinic for approximately 24 hours following each dose. Subjects may choose to have an optional lumbar puncture following the 3rd dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Men must practice a reliable method of birth control during study and for 2 weeks following study. Women must be non-fertile or post-menopausal.

Exclusion Criteria:

* Have serious or unstable illnesses as determined by the investigator.
* Have current or a history of asthma, or severe drug allergies or pollen allergy.
* Have used medications (except for calcium supplements or externally applied eye drops or antibiotics) within 30 days prior to dosing or are expected to use other medications during the study.
* Have had serious infectious disease affecting the brain within the preceding 5 years; or have known or existing evidence of serious infection.
* Have laboratory test values that are considered clinically significant as determined by the investigator.
* Have ECG abnormalities that are clinically significant.
* Have donated blood (a pint or more) or received an experimental drug within 30 days prior to dosing.
* Have a history of chronic alcohol or drug abuse within the past 2 years.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Pascuzzi, MD, Principal Investigator — IU Health Physicians - Neurology
Locations (1):
- IU Health Neuroscience Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CC100 (3 Single Doses): CC100 (3 single increasing doses by mouth). Dosing will occur every 2 to 7 days for a study duration of 5 to 15 days from the 1st dose.
  CC100
- CC100 (2 Single Doses) & Placebo(1 Dose): CC100 (2 single increasing doses by mouth) and placebo (1 single dose by mouth). Dosing will occur every 2 to 7 days for a study duration of 5 to 15 days from the 1st dose.
  CC100
  Placebo
Period: Overall Study
Arm/Group | CC100 (3 Single Doses) | CC100 (2 Single Doses) & Placebo(1 Dose)
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CC100 (3 Single Doses) | CC100 (2 Single Doses) & Placebo(1 Dose) | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Unsolicited Adverse Event Reports
Description: Safety and Tolerability assessed by arm/group and dose received measured by number of unsolicited AEs within a minimum of 24 hours after each dose.
Time Frame: Minimum of 24 hours after each dose.
Population: All 18 subjects analyzed, per protocol.
Measure: Number; unit: Unsolicited Adverse Event Reports
Arm/Group | CC100 (3 Single Doses) | CC100 (2 Single Doses) & Placebo(1 Dose)
Number analyzed (Participants) | 9 | 9
Unsolicited Adverse Event Reports | 3 | 4

2. Secondary Outcome: Pharmacokinetics (PK)
Description: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0.5, 1, 2, 3, 4, 5, 8, 12, 24 hrs post CC100
Population: 16 of 18 participants had data from drug level assays.The PK parameter analysis population included participants who received single CC100 dose(s) of 2, 5, 10, and/or 20 mg. Some PK parameters had fewer participants, if there were too few data points to analyze from a participant.
Measure: Mean (Standard Error); unit: hours
Groups:
- CC100 Single Doses: CC100: 2, 5, 10, and 20 mg/kg doses.
Arm/Group | CC100 Single Doses
Number analyzed (Participants) | 10
hours | 2.7 (2.3)

3. Secondary Outcome: Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0.5, 1, 2, 3, 4, 5, 8, 12, 24 hrs post CC100
Population: as for outcome 2
Measure: Mean (Standard Error); unit: hours
Arm/Group | CC100 Single Doses
Number analyzed (Participants) | 10
hours | 18.5 (14.2)

ADVERSE EVENTS:
Arm/Group | CC100 (3 Single Doses) | CC100 (2 Single Doses) & Placebo(1 Dose)
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 3/9 | 4/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CC100 (3 Single Doses) (N=9) | CC100 (2 Single Doses) & Placebo(1 Dose) (N=9)
Headache (Nervous system disorders) | 1 | 3
urinary tract infections (Infections and infestations) | 1 | 0
Fever (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No